CLINICAL TRIAL: NCT04148911
Title: An Open-Label, Phase IIIb, Single Arm, Multicenter Safety Study of Atezolizumab (Tecentriq) Plus Nab-Paclitaxel in the Treatment of Unresectable Locally Advanced or Metastatic Triple-Negative Breast Cancer
Brief Title: A Study of Atezolizumab Plus Nab-Paclitaxel in the Treatment of Unresectable Locally Advanced or Metastatic PD-L1-Positive Triple-Negative Breast Cancer
Acronym: EL1SSAR
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Hoffmann-La Roche (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: MO39874; 2019-002488-91 (EudraCT Number)
Record Dates: First submitted 2019-10-31; First posted 2019-11-04 (Actual); Results first posted 2025-12-26 (Actual); Last update posted 2025-12-26 (Actual); Status verified 2025-12

CONDITIONS: Triple-Negative Breast Cancer
MeSH Terms: conditions — Triple Negative Breast Neoplasms | interventions — atezolizumab; 130-nm albumin-bound paclitaxel; Albumin-Bound Paclitaxel

STUDY DESIGN:
Intervention Model Description: This is an open-label (non-blinded), single arm safety study in which all participants will receive atezolizumab in combination with nab-paclitaxel.
Masking Description: Open label, non-blinded
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (1):
- Atezolizumab plus Nab-Paclitaxel (Experimental): Participants will receive Atezolizumab via intravenous (IV) infusion on Days 1 and 15 of every 28-day cycle in combination with Nab-Paclitaxel on Days 1, 8, and 15 (individually selected by the investigator) until disease progression, or unacceptable toxicity, additionally until loss of clinical benefit as determined by the investigator or participant decision to discontinue treatment.
  Interventions: Drug: Atezolizumab; Drug: Nab-Paclitaxel

INTERVENTIONS:
Drug: Atezolizumab — Atezolizumab will be administered at a dose of 840 mg via IV infusion on Days 1 and 15 of every 28-day cycle. Day 15: Atezolizumab may be administered on Days 15-18 of each cycle.
  Other Names: Tecentriq
Drug: Nab-Paclitaxel — Nab-Paclitaxel will be administered at the 100 mg/m2 dose via IV infusion on Days 1, 8, and 15 of every 28-day cycle. Day 8: Nab-paclitaxel may be administered on Days 8-11 of each cycle. Day 15: Nab-paclitaxel may be administered on Days 15-18 of each cycle, on the same day with the atezolizumab infusion.
  Other Names: Abraxane

SUMMARY:
Study MO39874 is an open-label, Phase IIIb, single arm, global study conducted in participants with unresectable locally advanced or metastatic PD-L1-positive Triple-Negative Breast Cancer (TNBC) who have not received chemotherapy for their unresectable locally advanced or metastatic disease.

ELIGIBILITY:
Inclusion Criteria:

* Unresectable locally advanced or metastatic, histologically documented TNBC (negative for HER2 and ER and PgR)
* At least one specimen positive for PD-L1 status as determined by VENTANA PD-L1 SP142 IHC Assay
* No prior chemotherapy, experimental or targeted systemic therapy for unresectable locally advanced or metastatic TNBC
* Eastern Cooperative Oncology Group (ECOG) performance status of 0, 1 or 2
* Life expectancy ≥ 12 weeks
* Measurable disease, as defined by RECIST v1.1
* Adequate haematologic and end-organ function, defined by the following laboratory results obtained within 14 days prior to the initiation of study treatment
* Negative hepatitis B surface antigen (HBsAg) test at screening
* Negative total hepatitis B core antibody (HBcAb) test at screening, or positive HBcAb test followed by a negative hepatitis B virus (HBV) deoxyribonucleic acid (DNA) test at screening
* Negative hepatitis C virus (HCV) antibody test at screening, or positive HCV antibody test followed by a negative HCV ribonucleic acid (RNA) test at screening
* Patients with treated asymptomatic central nervous system (CNS) metastases are eligible, provided that all the following criteria are met: (a) The metastases are limited to the supratentorial region or cerebellum (b) No ongoing requirement for corticosteroids as therapy for CNS disease (c) No stereotactic radiation within 7 days or whole-brain radiation or neurosurgical resection within 2 weeks before the start of study treatment (d) Radiographic demonstration of interim stability between the completion of CNS-directed therapy and the screening imaging study.
* Patients with a history of autoimmune disease (Appendix 2) are allowed if controlled and on stable treatment (i.e., same treatment, same dose) for the last 12 weeks
* For women of childbearing potential: agreement to remain abstinent (refrain from heterosexual intercourse) or use contraceptive methods that result in a failure rate of < 1% per year, during the treatment period and for at least 5 months after the last dose of atezolizumab or 6 months after the last dose of nab-paclitaxel/paclitaxel, whichever is later. In addition, women must refrain from donating eggs during the same time period
* For men: agreement to remain abstinent (refrain from heterosexual intercourse) or use contraceptive measures and agreement to refrain from donating sperm
* Women who are not postmenopausal (≥ 12 months of non-therapy-induced amenorrhea) or surgically sterile must have a negative serum pregnancy test result within 14 days prior to initiation of study drug

Exclusion Criteria:

Cancer- Specific Exclusion Criteria:

* Spinal cord compression not definitively treated with surgery and/or radiation, or previously diagnosed and treated spinal cord compression without evidence that disease has been clinically stable for > 2 weeks prior to the first dose of study treatment (Cycle 1, Day 1).
* Leptomeningeal carcinomatosis or any symptomatic CNS metastases
* Uncontrolled symptomatic pleural effusion, pericardial effusion, or ascites
* Uncontrolled tumour-related pain
* Uncontrolled hypercalcemia (> 1.5 mmol/L ionized calcium or calcium > 12 mg/dL or corrected serum calcium > ULN) or symptomatic hypercalcemia requiring continued use of bisphosphonate therapy.
* Malignancies other than breast cancer within 5 years prior to the first dose of study treatment (Cycle 1, Day 1), with the exception of those with a negligible risk of metastasis or death and treated with expected curative outcome

General Medical Exclusion Criteria:

* Pregnancy or lactation
* Evidence of significant uncontrolled concomitant disease that could affect compliance with the protocol or interpretation of results, including significant liver disease
* Significant cardiovascular disease such as New York Heart Association (NYHA) cardiac disease (Class II or greater), myocardial infarction within 3 months prior to the first dose of study treatment (Cycle 1, Day 1), unstable arrhythmias, or unstable angina
* Severe infection within 4 weeks prior to the first dose of study treatment (Cycle 1, Day 1), including but not limited to hospitalization for complications of infection, bacteraemia, or severe pneumonia, or any active infection, that in the opinion of the investigator, could impact patient safety.
* Treatment with oral or IV antibiotics within 2 weeks prior to initiation of study treatment (Cycle 1, Day 1)
* Major surgical procedure within 28 days prior to the first dose of study treatment (Cycle 1, Day 1), or anticipation of the need for a major surgical procedure during the course of the study (other than diagnostic procedures)
* Treatment with investigational therapy within 4 weeks prior to Cycle 1, Day 1
* Known hypersensitivity to nab-paclitaxel or any of the excipients, when nab-paclitaxel is used as a backbone taxane
* Known hypersensitivity to paclitaxel or any of the excipients, when paclitaxel is used as a backbone taxane
* Positive human immunodeficiency virus (HIV) test at screening, unless the patient meets all of the following conditions: stable on anti-retroviral therapy, CD4 count ≥200/mL, undetectable viral load
* Any other disease, metabolic dysfunction, physical examination finding, or clinical laboratory finding that contraindicates the use of an investigational drug, may affect the interpretation of the results, or may render the patient at high risk from treatment complications

Exclusion Criteria Related to Atezolizumab:

* History of severe allergic, anaphylactic, or other hypersensitivity reactions to chimeric or humanized antibodies or fusion proteins
* Known hypersensitivity or allergy to biopharmaceuticals produced in Chinese hamster ovary cells or any component of the atezolizumab formulation
* Prior allogenic stem cell or solid organ transplantation
* History of idiopathic pulmonary fibrosis (including pneumonitis), drug-induced pneumonitis, organizing pneumonia (i.e., bronchiolitis obliterans, cryptogenic organizing pneumonia), or evidence of active pneumonitis on screening chest CT scan
* Current treatment with anti-viral therapy for HBV
* Active tuberculosis
* Receipt of a live, attenuated vaccine within 4 weeks prior to the first dose of study treatment (Cycle 1, Day 1), or anticipation that such a live, attenuated vaccine will be required during atezolizumab treatment or within 5 months following the final dose of atezolizumab
* Prior treatment with CD137 agonists or immune checkpoint blockade therapies (including anti-CTLA4 antibodies), except for anti-PD-1 or anti-PD-L1 antibodies.
* Treatment with systemic immunostimulatory agents (including but not limited to interferons or IL-2) within 4 weeks or five half-lives of the drug (whichever is longer) prior to the first dose of study treatment (Cycle 1, Day 1)
* Only in patients without autoimmune disease: Treatment with systemic corticosteroids or other systemic immunosuppressive medications (including but not limited to prednisone, dexamethasone, cyclophosphamide, azathioprine, methotrexate, thalidomide, and antitumour necrosis factor [TNF] agents) within 2 weeks prior to the first dose of study treatment (Cycle 1, Day 1), or anticipated requirement for systemic immunosuppressive medications during the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 184 (Actual)
Dates: Start 2019-12-10 (Actual); Primary Completion 2024-12-15 (Actual); Study Completion 2024-12-15 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Director — Hoffmann-La Roche
Locations (67):
- Argentina (3):
  - CEMIC, Buenos Aires
  - Sanatorio de la Mujer, Rosario
  - Organizacion Medica de Investigacion, San Nicolás
- Chile (2):
  - Instituto de Radiomedicina, IRAM, Santiago
  - Pontificia Universidad Catolica de Chile, Santiago
- Czechia (3):
  - Nemocnice AGEL Novy Jicin a.s., Nový Jičín
  - Fakultni Poliklinika Vseobecne Fakultni Niemocnice, Prague
  - Nemocnice na Bulovce, Prague
- France (6):
  - Institut de Cancérologie de Bourgogne, Dijon
  - Hôpital Franco-Britannique- Fondation Cognacq-Jay, Levallois-Perret
  - Centre Leon Berard, Lyon
  - Institut de cancerologie du Gard, Nîmes
  - Clinique Onco Des Dentellieres, Valenciennes
  - Departement Medecine, Villejuif
- Hungary (5):
  - Debreceni Egyetem Klinikai Kozpont, Debrecen
  - Bács-Kiskun Vármegyei Oktatókórház, Kecskemét
  - B-A-Z Vármegyei Központi Kórház és Egyetemi Oktatókórház, Miskolc
  - Komarom-Eszergom Varmegyei Szent Borbala Korhaz, Tatabánya
  - Zala Vármegyei Szent Rafael Kórház, Zalaegerszeg
- Italy (17):
  - Azienda Universitaria Magna Grecia, Catanzaro, Calabria
  - Azienda Ospedaliera San Giuseppe Moscati, Avellino, Campania
  - Policlinico Universitario Agostino Gemelli, Rome, Lazio
  - Irccs Ospedale San Raffaele, Milan, Lombardy
  - Istituto Europeo Di Oncologia, Milan, Lombardy
  - Ospedale San Gerardo, Monza, Lombardy
  - Fondazione IRCCS Policlinico San Matteo, Oncologia, Pavia, Lombardy
  - Ospedale Civile, Sassari, Sardinia
  - Ospedale Cannizzaro, Oncologia, Catania, Sicily
  - Fondazione del Piemonte per l?Oncologia (IRCCS), Candiolo, Trentino-Alto Adige
  - Ospedale Santa Chiara, Trento, Trentino-Alto Adige
  - Azienda ospedaliero-universitaria careggi, Sezione di radioterapia del dipartimento di fisiopatolo, Florence, Tuscany
  - Azienda Ospedaliero - Universitaria Pisana U.O. Oncologia Medica 2 Universitaria ? Polo Oncologico, Pisa, Tuscany
  - Nuovo Ospedale di Prato S. Stefano - Azienda USL Toscana Centro, Prato, Tuscany
  - Clinica Oncologica-Ospedali Riuniti Ancona, Torrette, Tuscany
  - USL Umbria 1 - Osp. Città di Castello, Città Di Castello (PG), Umbria
  - AULSS3 - Presidio di Mirano, Mirano (VE), Veneto
- Mexico (2):
  - Hospital de Oncología Siglo XXI, Mexico City, Mexico CITY (federal District)
  - Instituto Nacional de Cancerologia, Distrito Federal
- Peru (2):
  - Instituto Nacional de Enfermedades Neoplasicas, Lima
  - Hospital Nacional Cayetano Heredia, Lima
- Poland (4):
  - Szpital Specjalistyczny Podkarpacki O?rodek Onkologiczny, Brzozów
  - Szpital Wojewódzki im. Miko?aja Kopernika, Koszalin
  - Ars Medical Sp. z o. o., Pi?a
  - MRUKMED Lekarz Beata Madej-Mruk i Partner Spolka Partnerska Oddzial nr 1 w Rzeszowie, Rzeszów
- Portugal (6):
  - Hospital Garcia de Orta, Almada
  - IPO de Coimbra, Coimbra
  - IPO de Lisboa, Lisbon
  - Hospital de S. Francisco Xavier, Lisbon
  - Hospital Cuf Descobertas, Lisbon
  - IPO do Porto, Porto
- Romania (3):
  - Prof. Dr. I. Chiricuta Institute of Oncology, Cluj-Napoca
  - Centrul de Oncologie Sfantul Nectarie, Craiova
  - Centrul de Radioterapie AMETHYST, Floreşti
- Slovenia (2):
  - Institute of Oncology Ljubljana, Ljubljana
  - Univerzitetni klini?ni center Maribor, Maribor
- Spain (12):
  - Hospital General Universitario de Elche, Elche, Alicante
  - Corporacio Sanitaria Parc Tauli, Sabadell, Barcelona
  - Hospital Alvaro Cunqueiro, Vigo, Pontevedra
  - Hospital Univ. Central de Asturias, Oviedo, Principality of Asturias
  - Hospital de Basurto, Bilbao, Vizcaya
  - Hospital Universitario San Cecilio, Granada
  - Hospital Universitari Arnau de Vilanova de Lleida, Lleida
  - Hospital Lucus Augusti, Lugo
  - Hospital Universitario 12 de Octubre, Madrid
  - Hospital Clinico Universitario Virgen de la Victoria, Málaga
  - Hospital General Universitario J.M Morales Meseguer, Murcia
  - Hospital Clinico Universitario de Salamanca, Salamanca

IPD SHARING:
Plan to Share IPD: Yes
For eligible studies, qualified researchers may request access to individual patient level clinical data. See Roche's commitment to transparency of clinical study information here: https://go.roche.com/data_sharing
URL: https://www.clinicalstudydatarequest.com

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants with unresectable locally advanced or metastatic programmed death-ligand 1 (PD-L1)-positive Triple-Negative Breast Cancer (TNBC) took part in the study at 67 centers in 13 countries from 10 Dec 2019 to 15 Dec 2024.
Pre-assignment Details: Participants received atezolizumab in combination with nab-paclitaxel until disease progression (PD) or unacceptable toxicity or loss of clinical benefit. A total of 184 participants were enrolled in the study. However, two participants discontinued the study before receiving any treatment. Hence, participant flow data is presented for 182 participants. All protocol-specified assessments were completed as planned. Hence, this study was considered to be completed.
Groups:
- Atezolizumab + Nab-paclitaxel: Participants received atezolizumab 840 milligrams (mg) as intravenous (IV) infusion on Days 1 and 15 of each 28-day cycle along with nab-paclitaxel, 100 milligrams per square meter (mg/m^2) as IV infusion on Days 1, 8 and 15 of each 28-day cycle until PD, unacceptable toxicity, loss of clinical benefit or participant or investigator decision to discontinue treatment.
Period: Overall Study
Arm/Group | Atezolizumab + Nab-paclitaxel
Started | 182
Completed | 0
Not Completed | 182
Not completed — Death | 104
Not completed — Lost to Follow-up | 5
Not completed — Withdrawal by Subject | 17
Not completed — Study Ended by Sponsor | 56

BASELINE CHARACTERISTICS:
Population: Intent to Treat (ITT) population included all participants enrolled in the study. Out of the 184 enrolled participants, two participants discontinued and did not have any baseline data to analyze. Hence, data is presented for 182 participants.
Groups:
- Atezolizumab + Nab-paclitaxel: Participants received atezolizumab 840 mg as IV infusion on Days 1 and 15 of each 28-day cycle along with nab-paclitaxel, 100 mg/m^2 as IV infusion on Days 1, 8 and 15 of each 28-day cycle until PD, unacceptable toxicity, loss of clinical benefit or participant or investigator decision to discontinue treatment.
Arm/Group | Atezolizumab + Nab-paclitaxel
Number analyzed (Participants) | 182
Age, Continuous [Mean (Standard Deviation); unit: years] | 54.8 (12.2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 182
  Male | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 40
  Not Hispanic or Latino | 126
  Unknown or Not Reported | 16
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 17
  Asian | 1
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 1
  White | 146
  More than one race | 0
  Unknown or Not Reported | 17

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With Treatment-emergent Grade ≥3 Adverse Events (AEs)
Description: AE=untoward medical occurrence in participant administered a pharmaceutical product, regardless of causal attribution. AE=any unfavorable & unintended sign, symptom/disease temporally associated with the use of pharmaceutical product, whether/not considered related to it. Severity was graded per National Cancer Institute Common Terminology Criteria for Adverse Events version 5.0 (NCI CTCAE v5.0). Grade 1=Mild; asymptomatic/mild symptoms; clinical/diagnostic observations only; or intervention not indicated; Grade 2=Moderate; minimal, local/non-invasive intervention indicated; or limiting age-appropriate instrumental activities of daily living; Grade 3=Severe/medically significant, but not immediately life-threatening; hospitalization/prolongation of hospitalization indicated; disabling; or limiting self-care activities of daily living; Grade 4=Life-threatening consequences/urgent intervention indicated; Grade 5=Death related to AE. Percentages have been rounded off.
Time Frame: Up to 60 months
Population: Safety-evaluable population included all enrolled participants who had received at least one dose of any study treatment (atezolizumab/nab-paclitaxel).
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Atezolizumab + Nab-paclitaxel
Number analyzed (Participants) | 182
percentage of participants | 46.70 [39.29 to 54.23]

2. Primary Outcome: Percentage of Participants With Treatment-emergent Grade ≥2 Immune-mediated AEs (imAEs)
Description: AE=any untoward medical occurrence in a participant administered a pharmaceutical product, regardless of causal attribution. AE=any unfavorable and unintended sign, symptom/disease temporally associated with the use of a pharmaceutical product, whether/not considered related to it. Severity was graded according to NCI CTCAE v5.0. Grade 1=Mild; asymptomatic/mild symptoms; clinical/diagnostic observations only; or intervention not indicated; Grade 2=Moderate; minimal, local/non-invasive intervention indicated; or limiting age-appropriate instrumental activities of daily living (ADL); Grade 3=Severe/medically significant, but not immediately life-threatening; hospitalization/prolongation of hospitalization indicated; disabling; or limiting self-care ADL; Grade 4=Life-threatening consequences/urgent intervention indicated; Grade 5=Death related to AE. imAEs are events that resemble autoimmune diseases and are known side effects of immune checkpoint inhibitors.
Time Frame: Up to 60 months
Population: Safety-evaluable population included all enrolled participants who had received at least one dose of any study treatment (atezolizumab/nab-paclitaxel). Percentages have been rounded off.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Atezolizumab + Nab-paclitaxel
Number analyzed (Participants) | 182
percentage of participants | 12.09 [7.73 to 17.73]

3. Secondary Outcome: Percentage of Participants With All Treatment-emergent AEs
Description: An AE was any untoward medical occurrence in a participant administered a pharmaceutical product and which does not necessarily have to have a causal relationship with the treatment. An AE can therefore be any unfavorable and unintended sign (including abnormal laboratory values or abnormal clinical test results), symptoms, or disease temporally associated with the use of a pharmaceutical product, whether or not considered related to the PP. Percentages have been rounded off.
Time Frame: Up to 60 months
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Atezolizumab + Nab-paclitaxel
Number analyzed (Participants) | 182
percentage of participants | 95.60 [91.52 to 98.08]

4. Secondary Outcome: Percentage of Participants With All Treatment-emergent Serious Adverse Events (SAEs)
Description: An AE was any untoward medical occurrence in a participant administered a PP and which does not necessarily have to have a causal relationship with the treatment. An AE can therefore be any unfavorable and unintended sign (including abnormal laboratory values or abnormal clinical test results), symptoms, or disease temporally associated with the use of a pharmaceutical product, whether or not considered related to the PP. SAEs were defined as any AE that fulfilled any of the following criteria: fatal (resulted in death), life-threatening, required in-patient hospitalization or prolongation of existing hospitalization, resulted in persistent or significant disability/incapacity, was a congenital anomaly/ birth defect, was medically significant or required intervention to prevent any of the other outcomes listed here. Percentages have been rounded off.
Time Frame: Up to 60 months
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Atezolizumab + Nab-paclitaxel
Number analyzed (Participants) | 182
percentage of participants | 16.48 [11.41 to 22.69]

5. Secondary Outcome: Overall Survival (OS) in Safety-evaluable Population
Description: OS was defined as time from initiation of study treatment to death from any cause. OS was estimated using Kaplan-Meier (K-M) method.
Time Frame: Up to 60 months
Population: as for outcome 1
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Atezolizumab + Nab-paclitaxel
Number analyzed (Participants) | 182
months | 27.0 [22.0 to 33.8]

6. Secondary Outcome: OS in PD-L1-positive Population
Description: OS was defined as time from initiation of study treatment to death from any cause. OS was estimated using K-M method.
Time Frame: Up to 60 months
Population: PD-L1 positive population included all participants with centrally confirmed PD-L1 positive tumor status.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Atezolizumab + Nab-paclitaxel
Number analyzed (Participants) | 66
months | NA [29.4 to NA] — Median and upper limit of 95% CI were not estimable due to an insufficient number of participants with events.

7. Secondary Outcome: Progression Free Survival (PFS) in Safety-evaluable Population
Description: PFS was defined as the time from initiation of study treatment to the first occurrence of PD, as determined by the investigator according to Response Evaluation Criteria in Solid Tumors version 1.1 (RECIST v1.1), or death from any cause, whichever occurs first. PD was defined as at least a 20% increase in the sum of diameters of target lesions, taking as reference the smallest sum of diameters at prior timepoints (including baseline), and must also demonstrate an absolute increase of ≥ 5 millimeters (mm). PFS was estimated using K-M method.
Time Frame: Up to 60 months
Population: as for outcome 1
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Atezolizumab + Nab-paclitaxel
Number analyzed (Participants) | 182
months | 7.4 [5.6 to 10.6]

8. Secondary Outcome: PFS in PD-L1-positive Population
Description: PFS was defined as the time from initiation of study treatment to the first occurrence of PD, as determined by the investigator according to RECIST v1.1, or death from any cause, whichever occurs first. PD was defined as at least a 20% increase in the sum of diameters of target lesions, taking as reference the smallest sum of diameters at prior timepoints (including baseline), and must also demonstrate an absolute increase of ≥ 5 mm. PFS was estimated using K-M method.
Time Frame: Up to 60 months
Population: PD-L1 positive population included all participants with centrally confirmed PD-L1 positive tumor status.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Atezolizumab + Nab-paclitaxel
Number analyzed (Participants) | 66
months | 11.1 [7.4 to 16.8]

ADVERSE EVENTS:
Time Frame: Up to 60 months
Description: Safety-evaluable population included all enrolled participants who had received at least one dose of any study treatment (atezolizumab/nab-paclitaxel).
Arm/Group | Atezolizumab + Nab-paclitaxel
All-Cause Mortality (participants affected / at risk) | 104/182
Serious Adverse Events (participants affected / at risk) | 30/182
Other Adverse Events (participants affected / at risk) | 167/182
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Atezolizumab + Nab-paclitaxel (N=182)
Cardio-respiratory arrest (Cardiac disorders) | 1 (1)
Adrenal insufficiency (Endocrine disorders) | 1 (1)
Colitis (Gastrointestinal disorders) | 1 (1)
Diverticular perforation (Gastrointestinal disorders) | 1 (1)
Dysphagia (Gastrointestinal disorders) | 1 (1)
Chest pain (General disorders) | 1 (1)
Device related thrombosis (General disorders) | 1 (1)
Fatigue (General disorders) | 1 (1)
Oedema peripheral (General disorders) | 1 (1)
Pyrexia (General disorders) | 1 (1)
Hepatic failure (Hepatobiliary disorders) | 1 (1)
Device related sepsis (Infections and infestations) | 1 (1)
Infected skin ulcer (Infections and infestations) | 1 (1)
Myelitis (Infections and infestations) | 1 (1)
Pneumonia (Infections and infestations) | 1 (1)
Postoperative wound infection (Infections and infestations) | 2 (3)
Skin infection (Infections and infestations) | 1 (1)
Soft tissue infection (Infections and infestations) | 1 (1)
Subcutaneous abscess (Infections and infestations) | 1 (1)
Vascular device infection (Infections and infestations) | 1 (1)
Subdural haematoma (Injury, poisoning and procedural complications) | 1 (1)
Vascular access site inflammation (Injury, poisoning and procedural complications) | 1 (1)
Blood creatinine increased (Investigations) | 1 (1)
Transaminases increased (Investigations) | 1 (1)
White blood cell count decreased (Investigations) | 1 (1)
Dehydration (Metabolism and nutrition disorders) | 1 (1)
Electrolyte imbalance (Metabolism and nutrition disorders) | 1 (1)
Urinary tract obstruction (Renal and urinary disorders) | 1 (1)
Acute interstitial pneumonitis (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Bronchospasm (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 3 (3)
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Hypokalaemia (Metabolism and nutrition disorders) | 1 (1)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Atezolizumab + Nab-paclitaxel (N=182)
Anaemia (Blood and lymphatic system disorders) | 68 (160)
Leukopenia (Blood and lymphatic system disorders) | 27 (45)
Neutropenia (Blood and lymphatic system disorders) | 44 (118)
Hyperthyroidism (Endocrine disorders) | 14 (15)
Hypothyroidism (Endocrine disorders) | 34 (40)
Abdominal pain (Gastrointestinal disorders) | 12 (12)
Abdominal pain upper (Gastrointestinal disorders) | 12 (16)
Constipation (Gastrointestinal disorders) | 34 (42)
Diarrhoea (Gastrointestinal disorders) | 49 (73)
Dyspepsia (Gastrointestinal disorders) | 10 (16)
Nausea (Gastrointestinal disorders) | 50 (87)
Vomiting (Gastrointestinal disorders) | 22 (33)
Asthenia (General disorders) | 61 (106)
Fatigue (General disorders) | 34 (50)
Mucosal inflammation (General disorders) | 14 (21)
Oedema peripheral (General disorders) | 15 (25)
Pyrexia (General disorders) | 32 (42)
COVID-19 (Infections and infestations) | 28 (31)
Urinary tract infection (Infections and infestations) | 18 (21)
Alanine aminotransferase increased (Investigations) | 29 (53)
Blood alkaline phosphatase increased (Investigations) | 11 (18)
Blood lactate dehydrogenase increased (Investigations) | 13 (14)
Neutrophil count decreased (Investigations) | 15 (82)
White blood cell count decreased (Investigations) | 18 (60)
Decreased appetite (Metabolism and nutrition disorders) | 15 (19)
Hypokalaemia (Metabolism and nutrition disorders) | 10 (11)
Arthralgia (Musculoskeletal and connective tissue disorders) | 30 (37)
Back pain (Musculoskeletal and connective tissue disorders) | 19 (20)
Bone pain (Musculoskeletal and connective tissue disorders) | 10 (12)
Myalgia (Musculoskeletal and connective tissue disorders) | 30 (47)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 17 (17)
Dizziness (Nervous system disorders) | 13 (13)
Dysgeusia (Nervous system disorders) | 12 (13)
Headache (Nervous system disorders) | 24 (28)
Neuropathy peripheral (Nervous system disorders) | 24 (32)
Paraesthesia (Nervous system disorders) | 27 (33)
Insomnia (Psychiatric disorders) | 10 (12)
Breast pain (Reproductive system and breast disorders) | 10 (11)
Cough (Respiratory, thoracic and mediastinal disorders) | 19 (24)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 11 (12)
Alopecia (Skin and subcutaneous tissue disorders) | 72 (73)
Erythema (Skin and subcutaneous tissue disorders) | 14 (18)
Pruritus (Skin and subcutaneous tissue disorders) | 14 (18)
Rash (Skin and subcutaneous tissue disorders) | 22 (26)
Hypertension (Vascular disorders) | 10 (10)
Lymphoedema (Vascular disorders) | 12 (12)
Aspartate aminotransferase increased (Investigations) | 24 (32)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Study being conducted under this Agreement is part of the Overall Study. Investigator is free to publish in reputable journals or to present at professional conferences the results of the Study, but only after the first publication or presentation that involves the Overall Study. The Sponsor may request that Confidential Information be deleted and/or the publication be postponed in order to protect the Sponsor's intellectual property rights.

DOCUMENTS (2):
  • Study Protocol (2023-11-10): https://cdn.clinicaltrials.gov/large-docs/11/NCT04148911/Prot_000.pdf
  • Statistical Analysis Plan (2024-04-15): https://cdn.clinicaltrials.gov/large-docs/11/NCT04148911/SAP_001.pdf